CLINICAL TRIAL: NCT01188265
Title: Dextromethorphan Enhances the Therapeutic Efficacy of Valoproate in Bipolar Disorder Patients
Brief Title: Add-on Dextromethorphan in Bipolar Disorders
Acronym: DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-95-110
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid; Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Valproate & dextromethorphan 30 mg (Experimental): Valproate and dextromethorphan 30 mg per day
  Interventions: Drug: Valproate; Drug: Dextromethorphan 30 mg
- VPA & dextromethorphan 60 mg (Experimental): VPA & dextromethorphan 60 mg per day
  Interventions: Drug: Valproate; Drug: Dextromethorphan 60 mg per day
- VPA & Placebo (Active Comparator): VPA & placebo
  Interventions: Drug: Valproate; Drug: Placebo

INTERVENTIONS:
Drug: Valproate
Drug: Dextromethorphan 60 mg per day — VPA plus dextromethorphan 60 mg per day
  Arms: VPA & dextromethorphan 60 mg
Drug: Placebo — VPA plus placebo
  Arms: VPA & Placebo
Drug: Dextromethorphan 30 mg — VPA & Dextromethorphan 30 mg per day
  Arms: Valproate & dextromethorphan 30 mg

SUMMARY:
Dextromethorphan has been reported affording neuroprotection on dopaminergic neurons and having protective effect against inflammation-related neuron damage. These anti-inflammatory and neuroprotective effects of dextromethorphan would suggest potential clinical benefits of dextromethorphan add-on therapy to valproate for bipolar disorder patients. This hypothesis was based on the findings that the mood stabilizers have been reported to be neuroprotective through the release of neurotrophic factors such as GDNF from astroglia. Thus, the combination treatment of mood stabilizers and dextromethorphan might improve the therapeutic efficacy for bipolar disorder patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged ≧18 and ≦65 years.
2. A diagnosis of bipolar I or II disorder according to DSM-IV criteria made by a specialist in psychiatry.
3. A total of HDRS score at least 18 or YMRS score at least 14 at screen.
4. Signed informed consent by patient or legal representative
5. Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

1. Women of childbearing potential not using adequate contraception as per investigator judgment or not willing to comply with contraception for duration of study.
2. Females who are pregnant or nursing.
3. Patient has received dextromethorphan, or other selective cyclo- oxygenase 2 (Cox-2) inhibitors, or other anti-inflammatory medication within 1 week prior to first dose of double-blind medication.
4. Axis-I DSM-IV diagnosis other than bipolar I or II disorder.
5. Current evidence of an uncontrolled and/or clinically significant medical condition (e.g., cardiac, hepatic and renal failure), which in the judgments of the investigator, would compromise patient safety or preclude study participation.
6. History of intolerance to valproate or dextromethorphan or other Cox-2 inhibitors.
7. History of sensitivity reaction (e.g., urticaria, angioedema, bronchospasm, severe rhinitis, anaphylactic shock) precipitated by dextromethorphan.
8. Patient has received electroconvulsive therapy (ECT) within 4 weeks prior to first dose of doubleblind medication.
9. Diagnosis of or treatment for esophageal, gastric, pyloric channel, or duodenal ulceration or related complications (bleeding and/or perforation) within 30 days prior to receiving first dose of double-blind medication.
10. Inclusion in another bipolar disorder study or study for another indication with psychotropic's within the last 30 days prior to start of study.
11. Increase in total SGOT, SGPT, BUN and creatinine by more than 3X ULN (upper limit of normal).
12. History of idiopathic or drug-induced agranulocytosis.
13. Substance-related disorders within 6 months prior to study start, borderline personality disorder, schizophrenia, or other major psychiatric disorders as defined by DSM-IV criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Young's Mania Rating Scale (YMRS) | baseline, 1, 2, 4, 8 and 12 weeks
  The severity of current manic symptoms will be assessed by using the YMRS
Hamilton Depression Rating Scale (HDRS) | baseline, 1, 2, 4, 8 and 12 weeks
  The severity of depressive symptoms will be evaluated by HDRS

SECONDARY OUTCOMES:
blood samples | baseline, 1, 2, 4, 8 and 12 weeks
  The immune markers, cytokines will be measured at each time point to follow each patient's changes.
lipid profiles | baseline, after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Band Lu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Ru-Band Lu, Tainan, Taiwan